CLINICAL TRIAL: NCT01880333
Title: Phase 2/3 Study of the Modified Atkins Diet in Young Children With Refractory Epilepsy
Brief Title: Evaluation of the Modified Atkins Diet in Young Children With Refractory Epilepsy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Satinder Aneja, Director Professor, Lady Hardinge Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MADRE
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Refractory Epilepsy
Keywords: Refractory epilepsy; dietary therapy; non-pharmacological therapy; Modified Atkin Diet
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Children on Modified Atkin Diet (Experimental)
  Interventions: Other: Modified Atkin Diet

INTERVENTIONS:
Other: Modified Atkin Diet — Eligible children will be started on Modified Atkins diet with help of trained dietician. Carbohydrates intake will be restricted to 5 grams/ day in children<18 mo and 10grams/day in children 18mo- 3 years.Carbohydrate values of various food items will be explained in detail. Fats (e.g. cream, butter, oils, and ghee) will be encouraged. Proteins (cheese, fish, eggs, chicken, and soya products) will be unrestricted. Calcium and multivitamin supplementation will be done. Syrups will be restricted. Clear carbohydrates free fluids- will not be restricted. Medications will be changed to carbohydrate free preparations, wherever available. Diary of events will be recorded including seizure frequency and any adverse or positive effect. Urine ketones chart will be maintained.

SUMMARY:
The modified Atkins diet is a non-pharmacologic therapy for intractable childhood epilepsy that was designed to be a less restrictive alternative to the traditional ketogenic diet. This diet is started on an outpatient basis without a fast, allows unlimited protein and fat, and does not restrict calories or fluids. Modified Atkins diet is of special importance in resource constraint settings with paucity of trained dieticians. However, there is paucity published data on the use of the modified Atkins diet in refractory epilepsy in young children. This study aims to evaluate the efficacy and tolerability of the modified Atkins diet in refractory epilepsy in young children.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 9 months to 3 years.
2. Seizures persisting at least three per week for > 1 month despite the appropriate use of at least 2 Anti-epileptic drugs.

Exclusion Criteria:

1. Known or suspected inborn error of metabolism, as evidenced by: Clinical suspicion of metabolic disorder as evidenced by 2 or more of the following- a history of parental consanguinity, prior affected siblings, unexplained vomiting, intermittent worsening of symptoms, recurrent episodes of lethargy, altered sensorium, or ataxia, hepatosplenomegaly on examination And/ or 2 or more of the following biochemical abnormalities High blood ammonia (>80mmol/L), High arterial lactate (>2 mmol/L), metabolic acidosis (pH <7.2), hypoglycaemia (blood sugar <40 mg/dl), abnormal urinary aminoacidogram, presence of reducing sugars or ketones in urine, and positive results on urine neurometabolic screening tests.
2. Motivational or psychosocial issues in the family which would preclude compliance
3. Systemic illness- chronic hepatic, cardiac, renal or pulmonary disease
4. Severe acute malnutrition.

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children with > 50% seizure reduction at 3 months | After 3 months of diet initiation

SECONDARY OUTCOMES:
Frequency of adverse effects of the modified Atkins diet. | 3 months

OTHER OUTCOMES:
Proportion of children with seizure freedom at 3 months | 3 months
Percentage of children discontinuing diet before 3 months as per parenteral reports | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Satinder Aneja, MD, Principal Investigator — Kalawati Saran Children's Hospital, Lady Hardinge Medical College, New Delhi, India
Locations (1):
- Department of Pediatrics, Lady Hardinge Medical College and Associated Kalawati Saran Children's Hospital, New Delhi, National Capital Territory of Delhi, India